CLINICAL TRIAL: NCT05416359
Title: Phase I Clinical Trial of TQB3915 Tablets in Subjects With Advanced Malignant Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3915-I-01
Record Dates: First submitted 2022-06-09; First posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Advanced Malignant Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3915 tablets (Experimental): Take 300mg, 450mg, 600mg, 750mg, 900mg each time, once a day;Oral administration on an empty stomach, 28 days as a cycle. Duration of medication: Continue medication until disease progression or intolerable toxicity occurs.
  Interventions: Drug: TQB3915 tablets

INTERVENTIONS:
Drug: TQB3915 tablets — TQB3915 binds to estrogen receptors through covalent bonds, and blocks intracellular signal transmission by changing the conformation of ERα, thereby inhibiting the growth of tumor cells.

SUMMARY:
TQB3915 is a selective estrogen receptor covalent antagonist, by covalently binding to estrogen receptor, by changing the conformation of ERα, blocking intracellular signal transmission, thereby inhibiting the growth of tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* 1 Subjects voluntarily join the study and sign an informed consent form.
* 2 Age: 18-75 years old (when signing the informed consent form); Eastern Cooperative Oncology Group Performance status (ECOG PS) score: 0~1 points; Ected survival more than 3 months
* 3 Advanced malignant tumors clearly diagnosed by histology or cytology.
* 4 According to RECIST 1.1 criteria, it is confirmed that there is at least one measurable lesion;
* 5 The main organs are in good function,
* 6 Female subjects of childbearing age should agree to use contraceptive measures during the study period and within 6 months after the end of the study;

Exclusion Criteria:

* 1 Concomitant diseases and medical history:

  1. The previous pathological test was diagnosed as HER2-positive breast cancer;
  2. have inflammatory breast cancer;
  3. Other malignant tumors have occurred or are currently concurrently present within 3 years. The following two conditions were eligible for enrollment: other malignancies treated with a single surgery, achieving 5 years of disease-free survival (DFS); cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors [ Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor-infiltrating basement membrane)];
  4. There are multiple factors that affect oral medication (such as inability to swallow, acute and chronic diarrhea, and intestinal obstruction, etc.);
  5. Unresolved toxicity of CTC AE grade 1 and above due to any previous treatment, excluding alopecia;
  6. Subjects who have undergone major surgical treatment, significant traumatic injury, or are expected to undergo major surgery during the study period within 28 days prior to the first dose;
  7. wounds or fractures that have not healed for a long time;
  8. Those with a bleeding constitution; or suffering from clinically significant bleeding (such as hemoptysis), coagulation disorders, or being treated with antiplatelet/anticoagulants, blood transfusions or platelet transfusions;
  9. Have used a strong inhibitor or inducer of CYP3A within 2 weeks before taking the study drug for the first time;
  10. Arterial/venous thrombotic events, such as cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, occurred within 6 months before the first drug;
  11. Those who have a history of psychotropic substance abuse and cannot quit or have mental disorders;
  12. Subjects with any severe and/or uncontrolled disease, including:

      1. Poor blood pressure control (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg);
      2. Suffering from grade ≥2 myocardial ischemia or myocardial infarction, arrhythmia (including: QTc ≥450ms for males, QTc ≥470ms for females) and grade ≥2 congestive heart failure (New York Heart Association (NYHA) classification);
      3. Active or uncontrolled serious infection (≥CTC AE grade 2 infection);
      4. Liver cirrhosis; or active hepatitis: hepatitis B reference: HBsAg positive, and HBV DNA detection value exceeds the upper limit of normal; hepatitis C reference: HCV antibody positive, and HCV virus titer detection value exceeds the upper limit of normal; Note: Those who meet the entry conditions, subjects who are positive for hepatitis B surface antigen or core antibody, and subjects with hepatitis C, need to continue antiviral treatment to prevent virus activation;
      5. Active syphilis infection;
      6. Renal failure requiring hemodialysis or peritoneal dialysis;
      7. History of pulmonary interstitial fibrosis, drug-induced interstitial lung disease; or evidence of active pneumonia found on chest CT scan during screening;
      8. Those with a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
      9. Those who suffer from epilepsy and need treatment;
* 2 Tumor-related symptoms and treatment:

  1. Received surgery, chemotherapy, radiotherapy or other anti-cancer therapy within 4 weeks before the first dose (calculated from the end of the last treatment); those who have received local radiotherapy in the past can be included in the group if they meet the following conditions: The study treatment started more than 4 weeks (more than 2 weeks for brain radiotherapy); and the target lesions selected in this study were not in the radiotherapy area; or the target lesions were located in the radiotherapy area, but progress was confirmed;
  2. Received NMPA-approved Chinese patent medicines with anti-tumor indications in the drug instructions within 2 weeks before the first administration (including Compound Cantharidin Capsule, Kangai Injection, Kanglaite Capsule/Injection, Aidi Injection, Brucei Oil Injection /capsule, Xiaoaiping tablet/injection, cinobufacin capsule, etc.) treatment;
  3. Imaging (CT or MRI) shows that the tumor has invaded around important blood vessels or the investigator judges that the tumor is very likely to invade important blood vessels and cause fatal bleeding during the follow-up study;
  4. Uncontrolled pleural effusion, pericardial effusion or ascites that still requires repeated drainage (judgment by the investigator);
  5. Brain metastases, spinal cord compression, cancerous meningitis with clinical symptoms (unless asymptomatic, or treated and stable, no imaging evidence of new brain metastases or brain metastases expansion has been found for at least 2 weeks after treatment for brain metastases , and discontinued steroid or anticonvulsant therapy for at least 14 days prior to initiation of study treatment).
* 3 Study treatment related:

  1. Vaccination history of live attenuated vaccine within 28 days before the first dose or plan to receive live attenuated vaccine during the study period;
  2. Allergic constitution, or known allergy to the active ingredients or excipients of the study drug;
  3. Active autoimmune disease requiring systemic therapy (eg, use of disease-modifying drugs, corticosteroids, or immunosuppressants) within 2 years prior to initiation of study treatment; alternative therapy (eg, thyroxine, insulin, or adrenal or pituitary therapy) Physiological corticosteroids for insufficiency, etc.) are not considered systemic therapy;
  4. Diagnosed with immunodeficiency disease or are receiving systemic glucocorticoid therapy or any other systemic immunosuppressive therapy (dose >10mg/day prednisone or other equivalent therapeutic hormone), and still within 2 weeks before the start of study treatment in continued use;
  5. are using drugs known to prolong the QTc interval;
  6. is taking a drug known to cause sinus bradycardia.
* 4 Those who participated in clinical trials of other anti-tumor drugs within 4 weeks before enrollment or did not exceed 5 drug half-lives;
* 5 Any factors that increase the risk of QTc interval prolongation or risk of arrhythmia, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained occurrence in first-degree relatives younger than 40 years of age sudden death;
* 6 Any factors that may increase the risk of sinus bradycardia, such as hyperkalemia, hypothyroidism, etc.;
* 7 According to the judgment of the investigator, there are concomitant diseases that seriously endanger the safety of the subjects or affect the completion of the study, or subjects who are considered unsuitable for enrollment for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | up to 7 months
  The following adverse events related to the trial drug occurred within 1 treatment cycle (34 days) of the subject's first dose
Maximum Tolerated Dose (MTD) | up to 7 months
  The MTD was the previous dose at which the following toxicities occurred
Recommended Phase II Dose (RP2D) | up to 7 months
  To evaluate RP2D of TQB3915 Tablets in patients with advanced malignant tumors

SECONDARY OUTCOMES:
Adverse Events (AEs), Serious Adverse Events (SAEs) and Treatment-Related Adverse Events (TRAEs) | up to 18 months
  Incidence of all adverse events (AE), serious adverse events (SAE), and treatment-related adverse events (TEAEs)
Time to reach maximum(peak )plasma concentration following drug administration (Tmax) | up to 18 months
  To characterize the pharmacokinetics of TQB3915 by assessment of time to reach maximum plasma concentration after single dosing
Maximum (peak) plasma drug concentration (Cmax) | up to 18 months
  Cmax is the maximum plasma concentration of TQB3915.
Elimination half-life (t1/2) | up to 18 months
  t1/2 is time it takes for the blood concentration of TQB3915 to drop by half.
Area under the plasma concentration-time curve from time zero to infinity(AUC0-∞) | up to 18 months
  To characterize the pharmacokinetics of TQB3915 by assessment of area under the plasma concentration time curve from the first dose to infinity.
Area under the plasma concentration-time curve from time zero to time t (AUC0-t) | up to 18 months
  To characterize the pharmacokinetics of TQB3915 by assessment of area under the plasma concentration time curve from the first dose to a certain time point.
Apparent total clearance of the drug from plasma after oral administration (CL/F) | up to 18 months
  CL/F is total clearance rate for TQB3915.
Apparent volume of distribution（Vz/F） | up to 18 months
  Vz/F is the apparent distribution volume of TQB3915.
Maximum (peak) steady-state plasma drug concentration during during multiple-dose administration （Css,max） | up to 18 months
  Css,max is the steady state maximum concentration of TQB3915 .
Degree of fluctuation(DF) | up to 18 months
  DF is the volatility coefficient of TQB3915
Minimum steady-state plasma drug concentration during a dosage interval (Css,min) | up to 18 months
  Css,min is the minimum plasma concentration of TQB3915
Mean steady state plasma concentrations during a dosage interval (Css-av) | up to 18 months
  Css-av is the mean steady state plasma concentrations of TQB3915
Area under the steady-state plasma concentration-time curve(AUC0-τ) | up to 18 months
  AUC0-τis the area under the steady-state plasma concentration-time curve of TQB3915
Overall response rate (ORR) | up to 18 months
  Percentage of participants achieving complete response (CR) and partial response (PR).
Disease control rate（DCR） | up to 18 months
  Percentage of participants achieving CR and PR and stable disease (SD).
Clinical benefit rate (CBR) | up to 18 months
  Percentage of subjects who achieved complete remission (CR), partial remission (PR) and stable disease (SD) for at least 24 weeks
Duration of Response (DOR) | up to 18 months
  The period from the participants first achieving CR or PR to disease progression.
Progression-free survival (PFS) | up to 18 months
  PFS is defined as the time from the first treatment to the first disease progression or death from any cause
Overall survival (OS) | up to 18 months
  OS is defined as the time from the first administration to all-cause death.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Sun Yat-Sen University Cancer Canter, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - First Affiliated Hospital with Nanjin Medical University (Jiangsu Province Hospital), Nanjing, Jiangsu